CLINICAL TRIAL: NCT05740839
Title: High-Intensity Interval Exercise in Young Adult Survivors of Pediatric Brain Tumors: A Pilot Feasibility Study (HYPE)
Brief Title: High-Intensity Interval Exercise in Young Adult Survivors of Pediatric Brain Tumors: A Pilot Feasibility Study
Acronym: HYPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Stahl Family Charitable Foundation (Unknown); The Childhood Brain Tumor Foundation (Unknown); Pedals For Pediatrics (Unknown)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-505
Record Dates: First submitted 2023-02-02; First posted 2023-02-23 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Brain Tumor
Keywords: Pediatric Brain Tumor; Exercise Program; HIIT Program; Pediatric Brain Tumor Survivors
MeSH Terms: interventions — High-Intensity Interval Training; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT Exercise Program Group (Experimental): Participants will be randomly assigned to the HIIT exercise group and receive:
  * 3x weekly for 16 week home-based virtually supervised High-Intensity Interval Training.
  * 16-week self-directed exercise follow up period.
  * 3 On-site visits at Week 1, 18 and 34 for assement testing and completion of questionnaires
  Interventions: Behavioral: HIIT Exercise Program
- Control Group (Active Comparator): Participants will be randomly assigned to the HIIT waitlist control group and receive:
  * Daily usual activities
  * 2 On-site visits at Week 1, and 18 for assement testing and completion of questionnaires
  * Option to complete 16 week, 3x weekly HIIT exercise program after initial 16 week period.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: HIIT Exercise Program — Exercise program with stationary bike via the Zoom platform.
  Other Names: High-Intensity Interval Training
  Arms: HIIT Exercise Program Group
Behavioral: Control Group — Usual Activities
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine whether a 16-week virtual, home-based, high-intensity interval training (HIIT) exercise program will improve physical, cognitive, and emotional health among young adult survivors of pediatric brain tumors.

The names of the study interventions involved in this study are/is:

* High-Intensity Interval Training (HIIT)

DETAILED DESCRIPTION:
This is a Pilot/Feasibility, randomized control, research study that will compare an exercise group to a control group on physical, social, and overall quality of life needs of pediatric brain tumor survivors who are now young adults.

Participants will be randomized (selected at random) for two groups: HIIT program group will complete a 16-week intervention period followed by a 16-week period with no intervention and the waitlisted control group will complete a 16-week period and will perform their usual, daily activities followed by an optional 16-week period in which they can complete the HIIT program.

Research procedures include screening for eligibility, study treatment including in-clinic evaluations of fitness and strength, blood collection, at-home zoom exercise sessions, self-administered activity logs, and survey questionnaires.

Participation in this research study is expected to last about 8 months.

It is expected that about 30 people will take part in this research study.

The Stahl Family Charitable Foundation, Pedal 4 Pediatrics, and the Childhood Brain Tumor Foundation are supporting this research study by providing funding for the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study-related procedures.
* At time of study are a young adult, aged 18-39 years.
* Histologically diagnosed brain tumor during childhood (diagnosed ≤18 years).
* Are at least 2 years post tumor-directed therapy.
* The effects of exercise on the developing fetus are unknown. For this reason, women of child-bearing potential must agree to undergo a pregnancy test and to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.
* Medically cleared to participate in exercise by their referred physician or a certified clinical exercise physiologist.
* Are without medical conditions that could exacerbate with exercise, such as bone disease (excluding bone metastases) at imminent risk of fracture or uncontrolled cardiopulmonary or metabolic diseases.
* Speak English and/or Spanish.
* Currently participate in less than or equal to 60 minutes of moderate or vigorous structured exercise/week.
* Does not smoke or vape (no smoking/vaping during previous 12 months).
* Willing to travel to DFCI for necessary data collection.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Diagnosis of primary spinal cord tumor.
* Pre-existing medical conditions such as uncontrolled cardiopulmonary disease, or metabolic diseases that could exacerbate with exercise.
* Patients with active malignancies.
* Patients who are pregnant.
* Actively on a weight loss diet.
* Participate in more than 60 minutes of moderate or vigorous structured exercise/week.
* Currently smokes or vapes.
* Unable to travel to DFCI for necessary data collection.
* May not be able to comply with the safety monitoring requirements of the study in the opinion of the investigator.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Attendance of Exercise Sessions | From first exercise session to final exercise session, up to 16 weeks
  Defined as participant attendance of >= 70% of the 48 HIIT exercise sessions.
Completion in Minutes of Exercise Sessions | From first exercise session to final exercise session, up to 16 weeks
  Defined as participant completion of >= 70% of the 90 minutes of exercise per week
HIIT Compliance | From first exercise session to final exercise session, up to 16 weeks
  Defined as obtaining +-5W of target power output for >= 40 seconds of high intensity minute
Barriers to Exercise Adherence | From first exercise session to final exercise session, up to 16 weeks
  Assessed through the 17-item Barriers to Recruitment Participation Questionnaire (BRPQ), 1-5 scale with 1 denoted as strongly agree and 5 as strongly disagree.
Participant Burden | From first exercise session to final exercise session, up to 16 weeks
  Assessed through the Perceived Research Burden Assessment (PRBA), 1-5 scale with 1 denoted as strongly disagree and 5 as strongly agree.

SECONDARY OUTCOMES:
Cognition | : From baseline to post-intervention, up to 43 weeks
  An assortment of tests will be executed through the NIH toolbox to measure overall cognition.
Cardiorespiratory Fitness | From baseline to post-intervention, up to 43 weeks
  Assessed through the use of a VO2 max (or submaximal if equipment is unavailable) cycle exercise stress test (Parvo Medics TrueOne 2400; Sandy, UT, USA).
Muscular Strength | From baseline to post-intervention, up to 43 weeks
  10-repetition maximum will be used to assess muscular strength.
Body Composition | From baseline to post-intervention, up to 43 weeks
  Bioelectrical Impedance Analysis (BIA), and blood pressure as measured twice on both arms with a seated position with a minimum of 1-minute interval and the higher pressure will be recorded when there are differences.
  BIA: Assessed via bioelectrical impedance using a validated device (Tanita 780, Arlington Heights, IL). Participants will be asked to remove their shoes and socks after which height will be taken using a stadiometer they will then proceed to move to the BIA and stand still on the device while holding the handles with their hands at their sides. The device will estimate body fat using an algorithm based on their age, sex, height, and body weight.
Fatigue | From baseline to post-intervention, up to 43 weeks
  BFI: A questionnaire of scale ratings 0 - 10 that focuses on cancer-related fatigue and tiredness.
Psychosocial Health | From baseline to post-intervention, up to 43 weeks
  Assessed through the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire, which is comprised of 27 items with scale ratings validated to measure physical, emotional, social, and functional well-being of cancer patients and survivors
Quality of Sleep | From baseline to post-intervention, up to 43 weeks
  Assessed through the Pittsburg Sleep Quality Index (PSQI), which is used to measure 7 components of the quality and patterns of sleep in participants.
Dietary Assessment, ASA-24 | Up to 3 days
  Participants will be provided with a login to enter dietary data measured by an automated, online self-administered 24-hour assessment tool.
ActiGraph - Physical Activity Monitoring | From baseline to post-intervention, up to 27 weeks
  Participants will be provided with an accelerometer (ActiGraph, Pensacola, FL) to wear for seven days at baseline and post-intervention testing visits and will be instructed to wear the water-resistant accelerometer at all times except for when swimming or bathing. The device will record activity data and will be electronically transferred to a computer via USB cable at time of completion.
Exercise Tolerance | From baseline to week 16, up to 32 weeks
  Will be recorded using the Exercise-Induced Feeling Inventory (EIF). Based on a 0-4 scale, it assesses the participant's feeling state change(s) post-exercise and is also used for the assessment of self-motivation to adhere to an exercise regimen. Participants will be asked to complete the inventory before and after each exercise session.
Pain Index | From baseline to post-intervention, up to 43 weeks
  BPI: A 9 item questionnaire to evaluate the severity of pain and the impact of pain on the participant's daily functioning.
Hip and Waist Circumference | From baseline to post-intervention, up to 43 weeks
  Hip and waist circumference will be assessed and recorded in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu